CLINICAL TRIAL: NCT03097276
Title: Management of Patients With High C-reactive Protein After Scheduled Resection of Colorectal Cancer: Pilot Study
Brief Title: Management of Patients With High C-reactive Protein After Scheduled Resection of Colorectal Cancer
Acronym: GESPACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ORTEGA CGE 2016
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Colon and/or Rectal Resection With Anastomosis for Cancer
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients who underwent open decompression surgery (Other)
  Interventions: Procedure: blood sample; Radiation: CT scan

INTERVENTIONS:
Procedure: blood sample — blood sample will be collected
Radiation: CT scan — CT scan

SUMMARY:
Anastomotic fistula is the most feared complication after surgical resection of colorectal cancer (CCR). It occurs in 6 to 15% of patients. Beyond the risk of death in the immediate postoperative period, the pain that it induces, the resources required for its management, the need for stomata with a negative impact on patients' quality of life and the prolongation of hospitalization, it also has a now-recognized adverse effect on long-term survival.

The early detection of this complication may limit its impact. C-reactive protein (CRP) has proved to be an early, reliable marker of the onset of infectious complications of colorectal surgery.

However, the diagnostic procedure to implement in these patients is not at all codified, since this population concerned by systematic CRP assay in the postoperative period is very recent.

The procedures to implement in these patients so that they can obtain the maximal benefit of an early diagnosis have not yet been established. An algorithm for the proactive clinical management must be drawn up to be able to confirm or rule out the presence of a fistula as soon as a high level of CRP is detected, and to propose a quick treatment to ensure that patients benefit from this early diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 and older,
* with a CRP level > 140 mg/L at D3 or CRP > 125 mg/L at D4 following colon and/or rectal resection with anastomosis (protected or not by an upstream stoma)
* without clinical signs of severe peritonitis (fever, severe sepsis, generalized abdominal contracture)
* who have provided written informed consent.

Exclusion Criteria:

* patients who have undergone intraperitoneal chemotherapy in the context of the surgical treatment for peritoneal carcinomatosis
* patients with a diagnosis of another infection that could explain the high CRP level,
* patients who underwent eventration repair at the time of the colorectal resection
* patients with an obvious indication for revisit surgery
* persons without health insurance cover
* adults under guardianship
* pregnant or beast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
proportion of patients with total hospitalization of less than 15 days during the first postoperative month | 45 days

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Dijon, Dijon, France

REFERENCES:
- [Result] Gozalichvili D, Fournel I, Sow AK, Guiraud A, Moreno-Lopez N, Orry D, Facy O, Ortega-Deballon P. Management of patients with high C-reactive protein levels after elective colorectal surgery: Pilot study on a proactive diagnostic and therapeutic approach (GESPACE). J Visc Surg. 2024 Aug;161(4):237-243. doi: 10.1016/j.jviscsurg.2024.06.002. Epub 2024 Jun 21. PMID 38908988